CLINICAL TRIAL: NCT02298959
Title: A Phase 1 Trial of MK-3475 Plus Ziv-Aflibercept in Patients With Advanced Solid Tumors
Brief Title: Testing the PD-1 Antibody, MK3475, Given With Ziv-aflibercept in Patients With Advanced Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2014-01984; NCI-2014-01984 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 15-703; 9676 (Other: Dana-Farber - Harvard Cancer Center LAO); 9676 (Other: CTEP); U01CA062490 (NIH); UM1CA186644 (NIH); UM1CA186709 (NIH)
Record Dates: First submitted 2014-11-21; First posted 2014-11-24 (Estimated); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Clinical Stage IV Cutaneous Melanoma AJCC v8; Metastatic Colorectal Carcinoma; Metastatic Malignant Solid Neoplasm; Metastatic Melanoma; Metastatic Ovarian Carcinoma; Metastatic Renal Cell Carcinoma; Platinum-Resistant Ovarian Carcinoma; Recurrent Melanoma; Recurrent Renal Cell Carcinoma; Refractory Melanoma; Refractory Renal Cell Carcinoma; Sarcoma; Stage IV Colorectal Cancer AJCC v8; Stage IV Ovarian Cancer AJCC v8; Stage IV Renal Cell Cancer AJCC v8
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Melanoma; Ovarian Neoplasms; Carcinoma, Renal Cell; Sarcoma | interventions — Biopsy; Specimen Handling; pembrolizumab; aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (pembrolizumab and ziv-aflibercept) (Experimental): Patients receive pembrolizumab intravenously (IV) over approximately 30 minutes and ziv-aflibercept IV over 1-2 hours on day 1. Cycles repeat every 2 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients undergo CT scan, MRI, blood sample collection and tumor biopsy throughout the study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Elastography; Biological: Pembrolizumab; Biological: Ziv-Aflibercept

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo tumor biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Magnetic Resonance Elastography — Undergo MRI
  Other Names: MRE
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; GME 751; GME751; Keytruda; Lambrolizumab; MK 3475; MK-3475; MK3475; Pembrolizumab Biosimilar BCD-201; Pembrolizumab Biosimilar GME751; Pembrolizumab Biosimilar QL2107; Pembrolizumab Biosimilar RPH-075; Pembrolizumab Biosimilar SB27; QL2107; RPH 075; RPH-075; RPH075; SB 27; SB-27; SB27; SCH 900475; SCH-900475; SCH900475
Biological: Ziv-Aflibercept — Given IV
  Other Names: Aflibercept; Aflibercept beta; AVE0005; Eylea; Vascular Endothelial Growth Factor Trap; VEGF Trap; VEGF Trap R1R2; VEGF-Trap; Zaltrap

SUMMARY:
This phase I trial studies the side effects and best dose of ziv-aflibercept when given together with pembrolizumab in treating patients with solid tumors that that may have spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body (advanced). Ziv-afibercept works by decreasing blood and nutrient supply to the tumor, which may result in shrinking the tumor. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving ziv-aflibercept together with pembrolizumab may be a better treatment for patients with advanced solid tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the safety, tolerability and recommended phase II dosing for the combination of ziv-aflibercept plus MK-3475 (pembrolizumab) in patients with unresectable stage III or stage IV melanoma, renal cell cancer, ovarian cancer, colorectal cancer, or sarcoma.

SECONDARY OBJECTIVES:

I. To obtain preliminary estimates of progression-free survival at 6 months. II. To obtain preliminary estimates of the rate of 1-year overall survival. III. To obtain preliminary estimates of the response rate. IV. To obtain preliminary estimates of time to progression. V. To perform correlative sciences that provide information regarding the mechanisms of action for this combination treatment.

OUTLINE: This is a dose-escalation and dose expansion study of ziv-aflibercept.

Patients receive pembrolizumab intravenously (IV) over approximately 30 minutes and ziv-aflibercept IV over 1-2 hours on day 1. Cycles repeat every 2 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients undergo computed tomography (CT) scan, magnetic resonance imaging (MRI), blood sample collection and tumor biopsy throughout the study.

After completion of study treatment, patients are followed up for at least 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* In dose escalation, patients must have histologically or cytologically confirmed metastatic disease from any solid tumor (NOS 10029000). In dose expansion part 1, patients must have histologically or cytologically confirmed metastatic melanoma (10053571), renal cell carcinoma (NOS 10038485), ovarian cancer (NOS 10033272), or colorectal cancer (10009951,10038045). In dose expansion part 2, patients must have PD-1 resistant melanoma (10053571), PD-1 resistant renal cancer (NOS 10038485), or sarcoma (10061271)
* Renal cell patients must have had at least one prior vascular endothelial growth factor (VEGF) tyrosine kinase inhibitor (TKI)
* Ovarian cancer patients must be resistant to platinum therapy; therapy (i.e. within 6 months of last platinum therapy); patients who received greater than two prior platinum containing regimens will not be eligible
* Patients with colorectal cancer should have failed at least one oxaliplatin-containing regimen
* No more than two prior therapies for metastatic disease
* Age >= 18 years. Because no dosing or adverse event data are currently available on the use of MK-3475 in combination with ziv-aflibercept in patients < 18 years of age, children are excluded from this study, but will be eligible for future pediatric trials
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%)
* Estimated life expectancy of greater than 6 months
* Leukocytes >= 2,000/mcL (within 10 days of treatment initiation)
* Absolute neutrophil count >= 1,500/mcL (within 10 days of treatment initiation)
* Platelets >= 100,000/mcL (within 10 days of treatment initiation)
* Hemoglobin >= 9 g/dL OR >= 5.6 mmol/L (within 10 days of treatment initiation)
* Serum total bilirubin =< 1.5 X upper limit of normal (ULN) OR direct bilirubin =< ULN for patients with total bilirubin levels > 1.5 ULN (within 10 days of treatment initiation)
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X institutional ULN OR =< 5 X ULN for patients with liver metastases (within 10 days of treatment initiation)
* Serum creatinine =< 1.5 X ULN or measured or calculated creatinine clearance (CrCl) >= 60 mL/min for subject with creatinine levels > 1.5 X institutional ULN (glomerular filtration rate [GFR] can also be used in place of creatinine or CrCl); creatinine clearance should be calculated per institutional standard (within 10 days of treatment initiation)
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy not requiring laboratory monitoring as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants; therapeutic Coumadin is not acceptable (within 10 days of treatment initiation)
* Activated partial thromboplastin time (aPTT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy not requiring laboratory monitoring as long as PT or PTT is within therapeutic range of intended use of anticoagulants (within 10 days of treatment initiation)
* Urine protein-creatinine ratio (UPCR) =< 1 on spot urinalysis or protein =< 500 mg/24 hour urine
* Archival tissue must be available or newly obtained core or excisional biopsy of a tumor lesion
* Patients must have measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* The effects of MK-3475 and ziv-aflibercept on the developing human fetus are unknown; for this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; patients should continue contraceptive measures for 6 months from the last dose of all study medications
* Female patients of childbearing potential should have a negative urine or serum pregnancy test within 24 hours prior to receiving the first dose of study medication; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Female patients of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication; patients of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year
* Should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of MK 3475 and ziv-aflibercept administrations
* Ability to understand and the willingness to sign a written informed consent document
* Dose expansion part 2 PD-1/PD-L1 resistant or refractory melanoma and renal cell cancer only: subjects must have received prior immunotherapy with an anti-PD-1 or anti-PD-L1 containing regimen and must have progressive or recurrent disease after prior PD-1/PD-L1 directed therapy; primary resistance is determined at the time of initial restaging from initiation of treatment, as evidenced by progression by RECIST 1.1; acquired resistance would be a subject who had a best overall RECIST response of stable disease, partial response, or complete response confirmed radiographically by a second scan who subsequently developed progressive disease by RECIST 1.1 at any time thereafter
* Dose expansion part 2 sarcoma only: subjects must have received standard of care treatment

Exclusion Criteria:

* Patients who have had chemotherapy, targeted small molecule therapy, or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier

  * Note: patients with =< grade 2 neuropathy are an exception to this criterion and may qualify for the study
  * Note: if patients received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Patients who are currently participating in or have participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
* Has had a prior monoclonal antibody within 4 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events (AEs) due to agents administered more than 4 weeks earlier
* Has a known additional malignancy that is progressing or requires active treatment; exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy
* Lesions suspected to be at higher-risk for bleeding such as bowel involvement with tumor that invades into the bowel wall or involves the intraluminal component of bowel by imaging or direct visualization or central pulmonary lesions
* Ulcerated skin lesions
* Full anti-coagulant therapy Coumadin; patients may be receiving therapeutic Lovenox, Fragmin, or other heparin product that does not require laboratory monitoring
* Poorly-controlled hypertension as defined blood pressure (BP) > 150/100 mmHg, or systolic (S) BP > 180 mmHg when diastolic (D) BP < 90 mmHg, on at least 2 repeated determinations on separate days within 3 months prior to study enrollment
* Pregnant or nursing women
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* Patients with carcinomatous meningitis should also be excluded
* Patients with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least 3 months prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to MK-3475 and ziv-aflibercept
* Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents; patients with vitiligo or resolved childhood asthma/atopy would be an exception to this rule; patients that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study; patients with hypothyroidism stable on hormone replacement or Sjogren's syndrome will not be excluded from the study
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Dose escalation and dose expansion part 1 only: Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or ziv-aflibercept (prior treatment with bevacizumab is not an exclusion criteria)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, interstitial lung disease or active, non-infectious pneumonitis, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* If pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment; pregnant women are excluded from this study because MK-3475 is an agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with MK-3475, breastfeeding should be discontinued if the mother is treated with MK-3475; these potential risks may also apply to other agents used in this study; MK-3475 may have adverse effects on a fetus in utero; furthermore, it is not known if MK-3475 has transient adverse effects on the composition of sperm; patients are excluded from this study if pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Men and non-pregnant, non-breast-feeding women may be enrolled if they are willing to use 2 methods of birth control or are considered highly unlikely to conceive; highly unlikely to conceive is defined as 1) surgically sterilized, or 2) postmenopausal (a woman who is >= 45 years of age and has not had menses for greater than 2 years will be considered postmenopausal), or 3) not heterosexually active for the duration of the study; the two birth control methods can be barrier method or a barrier method plus a hormonal method to prevent pregnancy; patients should start using birth control from study visit 1 throughout the study period up to 120 days after the last dose of study therapy; the following are considered adequate barrier methods of contraception: diaphragm, condom (by the partner), copper intrauterine device, sponge, or spermicide; appropriate hormonal contraceptives will include any registered and marketed contraceptive agent that contains an estrogen and/or a progestational agent (including oral, subcutaneous, intrauterine, or intramuscular agents); patients should continue contraceptive measures for 6 months from the last dose of all study medications; patients should be informed that taking the study medication may involve unknown risks to the fetus (unborn baby) if pregnancy were to occur during the study; in order to participate in the study they must adhere to the contraception requirement (described above) for the duration of the study and during the follow-up period defined; if there is any question that a patient will not reliably comply with the requirements for contraception, that patient should not be entered into the study; pregnancy: If a patient inadvertently becomes pregnant while on treatment with MK-3475, the patient will immediately be removed from the study; the site will contact the patient at least monthly and document the patient's status until the pregnancy has been completed or terminated; the outcome of the pregnancy will be reported without delay and within 24 hours if the outcome is a serious adverse experience (e.g., death, abortion, congenital anomaly, or other disabling or life-threatening complication to the mother or newborn); the study investigator will make every effort to obtain permission to follow the outcome of the pregnancy and report the condition of the fetus or newborn; if a male patient impregnates his female partner the study personnel at the site must be informed immediately and the pregnancy reported and followed; it is unknown whether MK-3475 is excreted in human milk; since many drugs are excreted in human milk, and because of the potential for serious adverse reactions in the nursing infant, patients who are breast-feeding are not eligible for enrollment
* Patients who are human immunodeficiency virus (HIV) positive may participate IF they meet the following eligibility requirements:

  * They must be stable on their anti-retroviral regimen, and they must be healthy from an HIV perspective
  * They must have a cluster of differentiation (CD)4 count of greater than 250 cells/mcL
  * They must not be receiving prophylactic therapy for an opportunistic infection
* Has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)
* Has received a live vaccine within 30 days prior to the first dose of trial treatment
* History within 6 months prior to treatment of myocardial infarction, severe/unstable angina pectoris, coronary artery bypass graft (CABG), New York Heart Association (NYHA) class III or IV congestive heart failure (CHF), stroke or transient ischemic attack (TIA)
* History within 3 months prior to treatment of grade 3-4 gastrointestinal (GI) bleeding/hemorrhage, treatment resistant peptic ulcer disease, erosive esophagitis or gastritis, infectious or inflammatory bowel disease, diverticulitis, pulmonary embolus, or other uncontrolled thromboembolic event
* Patients who are less than 4 weeks post-operative (op) after major surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2015-04-08 (Actual); Primary Completion 2025-05-21 (Actual); Study Completion 2027-01-20 (Estimated)

PRIMARY OUTCOMES:
Recommended combination dose of ziv-aflibercept and pembrolizumab | 4 weeks
  Will be assessed by dose-limiting toxicities. Safety will be evaluated for all treated patients using the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0. All adverse events recorded during the trial will be summarized and presented by dose level. For patients enrolled in the dose expansion phase of the trial, adverse events summaries will also be summarized according to disease cohort. The proportion of patients with grade-3 or higher adverse events will be presented with 90% exact binomial confidence interval.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Between the date of first dose of trial therapy and the date of objectively documented disease progression or cessation of trial therapy, whichever occurs first, assessed up to 12 weeks
  The ORR will be the proportion of patients achieving complete or partial response as their best response to therapy. The analysis will be descriptive and will be used to assess for early indications of efficacy. Will be summarized by disease type and in the aggregate, if appropriate. ORR will be estimated and will be summarized with 90% confidence intervals estimated using exact binomial methods.
Progression-free survival | Time from start of trial treatment until objective disease progression (per RECIST) or death, whichever occurs first, assessed up to 6 months
  The analysis will be descriptive and will be used to assess for early indications of efficacy. Will be summarized by disease type and in the aggregate, if appropriate. Will be summarized using the product-limit method of Kaplan-Meier; 90% confidence intervals will be based on log(-log[outcome]) methodology.
Overall survival | Time from start of trial treatment to death from any cause, assessed up to 12 months
  The analysis will be descriptive and will be used to assess for early indications of efficacy. Will be summarized by disease type and in the aggregate, if appropriate. Will be summarized using the product-limit method of Kaplan-Meier; 90% confidence intervals will be based on log(-log[outcome]) methodology.
Time-to-progression | Time interval between the dates of the start of trial treatment and first documentation of progressive disease, assessed up to 12 weeks
  The analysis will be descriptive and will be used to assess for early indications of efficacy. Will be summarized by disease type and in the aggregate, if appropriate. Will be summarized using the product-limit method of Kaplan-Meier; 90% confidence intervals will be based on log(-log[outcome]) methodology.

OTHER OUTCOMES:
Phenotype changes in cell populations | Baseline to up to 12 weeks
  Will be assessed by flow cytometry. Will be determined as a function of treatment. Subpopulations of peripheral blood mononuclear cells will be isolated, including but not limited to dendritic cells, T cells, and B cells. These include regulatory and effector immune panels, naïve and memory CD4, CD8 and natural killer lymphocyte populations.
Tie-2 expressing monocytes | Up to 12 weeks
  Will be examined.
Changes in antigen specific responses to known melanoma antigen epitopes (melanoma antigen recognized by T cells 1, NY-ESO-1) | Baseline to up to 12 weeks
  Will be determined utilizing HLA-A20201 peptide system for antigen-presenting cells (including dendritic cell maturation and presentation) and targets.
Humoral and cellular immune responses | Up to 12 weeks
  Will be investigated by enzyme-linked immunosorbent assays, enzyme-linked immunospots, and cytotoxic T cell chromium release assays.
Effects on tumor vasculature and vascular active molecules | Up to 12 weeks
  Will investigate the effects on tumor vasculature and vascular active molecules as a function of treatment with the two-drug combination. Studies will include monitoring VEGF, basic fibroblast growth factor, and hepatocyte growth factor levels. Circulating endothelial cells and progenitors will be studied as a function of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Frank S Hodi, Principal Investigator — Dana-Farber - Harvard Cancer Center LAO
Locations (9):
- United States (7):
  - Moffitt Cancer Center-International Plaza, Tampa, Florida
  - Moffitt Cancer Center - McKinley Campus, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - National Cancer Institute Developmental Therapeutics Clinic, Bethesda, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
- Canada (2):
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Baginska J, Nau A, Gomez Diaz I, Giobbie-Hurder A, Weirather J, Vergara J, Abrecht C, Hallisey M, Dennis J, Severgnini M, Huezo J, Marciello I, Rahma O, Manos M, Brohl AS, Bedard PL, Renouf DJ, Sharon E, Streicher H, Ott PA, Buchbinder EI, Hodi FS. Ziv-aflibercept plus pembrolizumab in patients with advanced melanoma resistant to anti-PD-1 treatment. Cancer Immunol Immunother. 2024 Jan 18;73(1):17. doi: 10.1007/s00262-023-03593-2. PMID 38236249
- [Derived] Rahma OE, Tyan K, Giobbie-Hurder A, Brohl AS, Bedard PL, Renouf DJ, Sharon E, Streicher H, Hathaway E, Cunningham R, Manos M, Severgnini M, Rodig S, Stephen Hodi F. Phase IB study of ziv-aflibercept plus pembrolizumab in patients with advanced solid tumors. J Immunother Cancer. 2022 Mar;10(3):e003569. doi: 10.1136/jitc-2021-003569. PMID 35264434